CLINICAL TRIAL: NCT01481103
Title: Integrating Acupuncture Into the Management of Migraines: A Randomized, Comparative Trial
Brief Title: Integrating Acupuncture Into the Management of Migraines
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI cited personal reasons
Sponsor: National University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUHS H1009
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Migraine Headache
Keywords: Over the counter medication; Acupuncture
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture group (Active Comparator): Participants will keep a headache diary for 4weeks and then attend eight weekly acupuncture sessions. Acupuncture will be done by a licensed acupuncturist and will last approximately 25 minutes. Following the acupuncture sessions, participants will keep a headache diary for an additional 4 weeks
  Interventions: Procedure: Acupuncture
- Control group (No Intervention): participants will be asked to maintain a daily diary of headache occurrences and OTC medication use for 16 weeks.

INTERVENTIONS:
Procedure: Acupuncture — participants will receive 8 weekly acupuncture sessions. Acupuncture will be performed by a licensed acupuncturist. Each session will last approximately 25 minutes.
  Arms: Acupuncture group

SUMMARY:
This research is being done to study the effect of incorporating acupuncture into the management of migraines. The primary aim is to determine in a randomized, controlled study whether individuals experiencing migraines have fewer occurrences and less intense migraines when acupuncture is integrated with nonprescription pharmacological treatment. Nonprescription pharmacological treatment in this study refers to the use of the following over the counter medications: Aspirin, Ibuprofen, Naproxen, Acetaminophen (with or without caffeine). Aspirin, Ibuprofen, and Naproxen are members of a class of drugs known as non-steroidal anti-inflammatory drugs or NSAIDs.

DETAILED DESCRIPTION:
70 men and women between the ages of 18-65 diagnosed with migraines by a medical doctor. Participants must be using only nonprescription medication to treat their head pain.

Once initial eligibility has been determined and informed consent obtained, a Traditional Chinese Medicine (TCM) differential diagnosis will be carried out to determine the underlying cause of the migraines experienced by the participant. If the migraines are due to Liver Qi stagnation with Liver Yang rising they will be eligible for participation in the study. Eligible participants will be randomly assigned to one of two groups: Group 1 will continue taking their current nonprescription migraine medication as needed and will receive acupuncture once a week for 8 weeks. Group 2 will continue with their current nonprescription migraine medication as needed but will not receive acupuncture. The same set of predetermined acupuncture points will be used at each session.

All participants will complete a daily headache and medication use diary for four weeks on two separate occasions. In addition all participants will complete the Headache Impact Test (HIT-6) survey on three separate occasions.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with or without aura according to the International Headache Society classification and diagnosed by a Medical Doctor.
* Subjects are required to have between 2 and 12 migraines but no more than 15 headache days (migraine or nonmigraine) per 28 days during the prospective baseline phase. A headache day is defined as a calendar day during which the patient experienced headache for at least 30 minutes.
* Taking a nonprescription medication for the migraine pain. More specifically Aspirin, Ibuprofen, Naproxen, and/or Acetaminophen (with or without caffeine).
* Age between 18 and 65 years.
* A history of migraine for at least 12 months.
* Completed at least 75% of the baseline headache diary.
* Completion of written informed consent.

Exclusion Criteria:

* Onset of headache disorder less than 12 months prior to age 50.
* Pregnancy or planning to get pregnant while participating in the study.
* Malignancy; cluster headache (IHS code 3); sinus headaches.
* Suspicion that headache disorder has specific etiology (IHS code 5-11); cranial neuralgias (IHS code12)
* Acupuncture treatment in the previous 12 months.
* Taking a prescription medication for the migraine pain.
* Subject plans to receive acupuncture for another medical condition while participating in the study.
* Systemic disorder or illness, including serious psychiatric illness.
* Failure to fulfill baseline information.
* Failure to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number and intensity of migraine headaches | 16 weeks
  Participants will be asked to maintain a daily diary of headache occurrences and medication use for 4 weeks prior to intervention and 4 weeks after intervention

SECONDARY OUTCOMES:
Medication consumed | 16 weeks
  Participants will be asked to maintain a daily diary of headache occurrences and medication use for 4 weeks prior to intervention and 4 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Miller, LAc, PT, Principal Investigator — National University of Health Sciences; Hui Yan Cai, LAc, PhD, Study Director — National University of Health Sciences
Locations (1):
- Serenity Acupuncture and Oriental Medicine, Oak Park, Illinois, United States